CLINICAL TRIAL: NCT00000171
Title: Study of Melatonin: Sleep Problems in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0006; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Alzheimer Disease; Dyssomnias
Keywords: Alzheimer's disease; Sleep disorders; Melatonin
MeSH Terms: conditions — Alzheimer Disease; Dyssomnias; Sleep Wake Disorders | interventions — Melatonin

INTERVENTIONS:
Drug: Melatonin

SUMMARY:
This protocol is a multicenter clinical trial of melatonin for sleep disturbances associated with Alzheimer's disease (AD). Frequent nocturnal awakening is a common behavioral symptom of AD. Nighttime wandering and agitated behavior may result in injuries and sleep disruption for caregivers. Alternatives are sorely needed to the currently available sleep medications that have marginal efficacy and serious side effects. Melatonin is a naturally occurring hormone secreted by the pineal gland. It has soporific effects with oral administration and is well tolerated. It enhances sleep in normal older people. Melatonin also may help sleep disturbances associated with AD; however, this remains to be proven.

DETAILED DESCRIPTION:
In Alzheimer's disease , sleep disruption is one of the most common behavioral problems, occurring in 45 percent of patients. These nocturnal awakenings and agitation lead to considerable burden for caregivers and frequently lead families to the decision of nursing home placement. The proposed study is a randomized, double blind, parallel group, placebo controlled, clinical trial. Placebo will be compared with two doses of melatonin: a 2.5 mg, slow- release preparation and a 10 mg immediate release preparation. One hundred and fifty community-residing AD patients with disrupted sleep will be recruited. Included subjects will meet NINCDS-ADRDA criteria for probable AD. Prior to study entry, disrupted sleep will be documented by clinical history and by 1 to 2 weeks of recording using wrist activity monitors. The treatment period will last 8 weeks. Rest/activity patterns will be recorded by wrist activity monitors. The primary outcome measure will be the change in nocturnal sleep time from baseline to the end of the treatment phase.

Other outcomes also will be examined, including the time awake after sleep onset, sleep latency, sleep efficiency, daytime agitation, and changes in cognition. The relative effectiveness of high and low dose melatonin will be assessed. Adverse events and side effects will be compared by treatment. This study should provide the data necessary to determine whether melatonin is a safe and effective treatment for disrupted sleep associated with AD.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet NINCDS-ADRDA criteria for probable Alzheimer's disease (AD). Patients must have disrupted sleep, documented by clinical history and by 1 to 2 weeks of recording using wrist activity monitors.
* A diagnosis of probable AD.
* MMSE score 0-26.
* Hachinski Ischemia Scale score less than or equal to 4.
* A 2-week history of two or more sleep disorder behaviors, occurring at least once weekly, as reported by the caregiver on the Sleep Disorder Inventory.
* CT or MRI since the onset of memory problems showing no more than one lacunar infarct in a non-strategic area and no clinical events suggestive of stroke or other intracranial disease since the CT or MRI.
* Physically acceptable for study as confirmed by medical history and exam, clinical laboratory results, and EKG.
* Actigraph evidence of a mean nocturnal sleep time of less than 7 hours per night (at least 5 nights of complete actigraph data must be collected over a single week.
* Stable home situation with no planned move during the 13-week investigational period.
* Residing with responsible spouse, family member, or professional caregiver who is present during the night and will agree to assume the role of the principal caregiver for the 13-week protocol, including arranging transport for the patient to and from the investigators' clinic, answering questions regarding the patient's condition, and assuming responsibility for medication and actigraph procedures.
* Ability to ingest oral medication and participate in all scheduled evaluations.
* Six grades of education or work history sufficient to exclude mental retardation.
* 55 years of age or older.
* Hamilton Depression Rating Scale score of 15 or less.
* Stable medication (dose and type) for non-excluded concurrent medical conditions for 4 weeks prior to the screening visit.

Exclusion Criteria:

* Sleep disturbance is acute (within the last 2 weeks).
* Sleep disturbance is associated with an acute illness with delirium.
* Clinically significant movement disorder that would interfere with the actigraph readings.
* Not having a mobile upper extremity to which to attach an actigraph.
* Severe agitation.
* Pain syndrome affecting sleep.
* Unstable medical condition.
* Use of investigational or unapproved medications within 4 weeks of the screening visit.
* Patient unwilling to maintain caffeine abstinence after 2:00 pm for the duration of the protocol.
* Patient unwilling to comply with the maximum limit of two alcoholic drinks per day, and only one alcoholic drink after 6:00 pm for the duration of the protocol.
* Use of melatonin within 2 weeks of screening visit.
* Clinically significant abnormal laboratory findings that have not been approved by the Project Director.
* Residing in a facility without a consistent caregiver present during the night who can function as the primary informant.
* Caregiver deemed too unreliable to supervise the wearing of the actigraph, to maintain the sleep diary, or to bring the patient to the scheduled visits.
* Autoimmune disease, such as rheumatoid arthritis and polymyalgia rheumatica.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Cliff Singer, M.D., Study Director — Oregon Health and Science University
Locations (31):
- United States (31):
  - University of Arizona, Tucson, Arizona
  - University of California Irvine Institute for Brain Aging and Dementia, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Yale University, Alzheimer's Disease ResearchUnit, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mount Sinai (Miami), Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta VA Medical Center, Augusta, Georgia
  - Southern Illinois University, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic at Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Pawtucket, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Singer C, Tractenberg RE, Kaye J, Schafer K, Gamst A, Grundman M, Thomas R, Thal LJ; Alzheimer's Disease Cooperative Study. A multicenter, placebo-controlled trial of melatonin for sleep disturbance in Alzheimer's disease. Sleep. 2003 Nov 1;26(7):893-901. doi: 10.1093/sleep/26.7.893. PMID 14655926
- [Derived] McCleery J, Sharpley AL. Pharmacotherapies for sleep disturbances in dementia. Cochrane Database Syst Rev. 2020 Nov 15;11(11):CD009178. doi: 10.1002/14651858.CD009178.pub4. PMID 33189083
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging (NIA). — http://www.alzheimers.org